CLINICAL TRIAL: NCT04300816
Title: Efficacy of a Psychosocial Intervention to Improve Ability to Cope With Uncertainty in MS
Brief Title: Coping and Adjusting to Living With Multiple Sclerosis
Acronym: CALMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Ivan Molton, Professor, School of Medicine: Rehabilitation Medicine: Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00007984
Record Dates: First submitted 2020-03-04; First posted 2020-03-09 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: 3- arm randomized clinical trial. Arms: (1) CBT for uncertainty tolerance, (2) traditional CBT, (3) treatment as usual
Who Masked: Outcomes Assessor
Masking Description: Research manager will be blinded for this trial. Research coordinator and investigator will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT-UT (Experimental): Seven telephone-based sessions of cognitive behavioral therapy for uncertainty tolerance (CBT-UT) delivered over seven weeks.
  Interventions: Behavioral: CBT for Uncertainty Tolerance
- tCBT (Active Comparator): Seven telephone-based sessions of traditional cognitive behavioral therapy (tCBT) delivered over seven weeks.
  Interventions: Behavioral: Traditional CBT
- TAU (No Intervention): Participant continues with their lives as they normally would.

INTERVENTIONS:
Behavioral: CBT for Uncertainty Tolerance — Participants work one-on-one with an interventionist. Treatment sessions focus on understanding the difference between the controllable and uncontrollable aspects of MS, ability to tolerate not knowing exactly what the future will hold, setting personal goals for what "accepting" what MS will look like, and finding ways to live in conjunction with personal values despite the MS diagnosis.
  Other Names: CBT-UT
  Arms: CBT-UT
Behavioral: Traditional CBT — Participants work one-on-one with an interventionist. Treatment sessions focus on goal setting, positive activities, identifying and challenging unhelpful thoughts, and bolstering social support.
  Other Names: tCBT
  Arms: tCBT

SUMMARY:
The purpose of this project is to test a brief, telephone-based psychological intervention, CBT-UT, to improve the ability to tolerate uncertainty-and thereby to reduce distress-in people with a recent diagnosis of Multiple Sclerosis (MS). There are three treatment arms for this study. Participants will receive either (1) CBT for Uncertainty Tolerance, (2) Traditional CBT, or (3) treatment as usual.

DETAILED DESCRIPTION:
Despite substantial improvements in diagnosis and treatment, Multiple Sclerosis (MS) remains an unpredictable disease. Although some physicians can make some predictions about expected progression, the variable course of exacerbations makes it almost impossible to predict how MS will develop or affect function over time. As a result, people with MS must learn to live in a state of chronic uncertainty and the ability to tolerate and cope with this kind of uncertainty is central to quality of life with MS. Individuals who require certainty about the future and are not able to tolerate ambiguity are said to be high in a personality trait known as intolerance of uncertainty (IU). There is a significant gap in MS clinical intervention that necessitates attention. An intervention that specifically targets IU, is developed for people recently diagnosed with MS, and can be provided remotely via telehealth can make a significant impact for this population. Study aims include: (1) to determine the efficacy of CBT-UT relative to traditional cognitive behavioral therapy (tCBT) or treatment as usual (TAU) in people diagnosed with MS in the past 3 years; and (2) To increase our understanding of the mechanisms underlying the intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* MS diagnosis using revised McDonald Criteria
* Able to read, speak, and understand English
* At least mild psychological distress evidenced by (1) a score of 20 or higher on the Kessler Psychological Distress Scale OR (2) a score greater than or equal to 5 on the Perceived Stress Scale.

Exclusion Criteria:

* Severe cognitive impairment defined as one or more error on the Six-Item Screener
* Psychiatric condition or symptoms that would interfere with participation, specifically (1) current, active suicidal ideation with current intent to harm oneself, (2) current psychosis, or (3) current mania.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Questionnaire: Level of MS Acceptance as measured by the Acceptance of Chronic Health Conditions, MS Version Questionnaire. | 6 Months
  This is a self-reported measure of perceived MS Acceptance. Greater scores represent greater MS Acceptance.
Questionnaire: Level of anxiety as measured by the Global Anxiety Disorder-7 scale (GAD-7). | 6 Months
  This is a self-reported measure of perceived anxiety. Greater scores represent greater levels of anxiety.
Questionnaire: Level of depression as measured by the Patient Health Questionnaire (PHQ-9). | 6 Months
  This is a self-reported measure of perceived depression. Greater scores represent greater levels of depression.

SECONDARY OUTCOMES:
Demographic: MS Progression Type. Measured by self-reported type of MS. | Baseline
  This is a self-reported demographic question. Options include: Relapsing-Remitting, Primary-Progressive, Secondary-Progressive, Progressive-Relapsing, and Don't Know.
Demographic: Biological Sex. Measured by self-report. | Baseline
  This is a self-reported demographic question. Options include: Male, Female, Transgender, and If not listed explain.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Molton, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators propose to make available to interested researchers a data file (de-identified to remove any variables from which it would be possible to identify any individual participant) any data used in a published article, at the time that it is accepted for publication. That is, at the request of an outside researcher, the investigators will create and share a data file that includes all of the variables used in the published article and a list of the variables in the data file (along with their variable labels). Any investigators who request these data will receive (1) a copy of the published article (which will describe the source of the data); (2) the variable list/variable labels; and (3) a data set.
Time Frame: Data will become available after the main study results are published.
Access Criteria: Although any shared data will be stripped of identifiers prior to release, given the very specific nature of the study sample (individuals who have had a recent diagnosis of MS) it is possible that those who access this data could potentially identify subjects with unusual characteristics or combinations of unusual characteristics. Therefore, the investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.